CLINICAL TRIAL: NCT00216814
Title: Intravesically Administered BCG May Have Antiangiogenic Effects on Urinary Concentrations of Basic Fibroblast Growth Factor ( bFGF), Vascular Endothelial Growth Factor (VEGF) and Interleukin (IL-8)
Brief Title: Antiangiogenic Effects of BCG on Urinary Concentration of Angiogenic Factors
Status: Terminated | Type: Observational
Why Stopped: No funding and data was not appropriate to consider continuing.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: R-03-275; 10050E
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-01

CONDITIONS: Bladder Cancer
Keywords: antiangiogenic effects of bcg treatment and prognosis
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To determine if there is an association between basic fibroblast growth factor,vascular endothelial growth factor, and interleukin levels and a patients response to BCG treatment ( as standard treatment)in the urine of patients with superficial TCC. To determine if the levels of these angiogenic factors can predict response to BCG, disease recurrence, progression risk factors.

DETAILED DESCRIPTION:
200 patients that are candidates for intravesical BCG therapy and 20 control patients with no history of malignancy will be enrolled. The study group wol;; be asked to provide a urine sample just prior to receiving their first BCG treatment(week # 1) and just prior to receiving their last (week # 6) BCG treatment. The control patients will provide one urine sample only. Samples will be analysed by enzyme-linked immunosorbant assay(ELISA). clinical data will be reviewed on tumor stage and grade prior to BCG, timme to recurrence, tumor stage and grade of recurrence, time to disease progression and death, cause of death and total follow-up time.

ELIGIBILITY:
Inclusion Criteria:

200 study group 1. Must be a candidate for BCG therapy. 20 control group 1. No history of malignancy.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bladder cancer that are receiving treatment with BCG.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2003-10; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Izawa, MD, FRCSC, Principal Investigator — LHRI
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada